CLINICAL TRIAL: NCT05711264
Title: Presence of Circulating CD4+CD28 Null T Helper Lymphocytes in Patients With Autoimmune Hemolytic Anemia.
Brief Title: Presence of Circulating Cluster of Differentiation 4 Positive 28 Null T Helper Lymphocytes(CD4+CD28-) in Patients With Autoimmune Hemolytic Anemia.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Ehab Salah Eldin, Resident in clinical pathology department, Assiut University
Other Study IDs: CD4+CD28- Lymphocyte IN AIHA
Record Dates: First submitted 2023-01-13; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Autoimmune Hemolytic Anemia
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Study the presence of circulating CD4+/CD28 null T lymphocytes in AIHA either Idiopathic or Secondary.
2. Role of CD4+/CD28 null T lymphocytes in monitoring response to therapy in AIHA.

DETAILED DESCRIPTION:
Autoimmune hemolytic anemia (AIHA) has always been considered the simplest and most scholastic example of antibody-mediated autoimmune disease.It has been identified as a greatly heterogeneous disease, due to several immunological mechanisms involved beyond antibodies, complement and antibody-dependent cell-mediated cytotoxicity (ADCC). AIHAs may be Idiopathic of unknown cause Secondary associated with several conditions : (lymphoproliferative, autoimmune , infectious diseases, immunodeficiencies, solid tumors, transplants, and drugs).Several subsets of T and B lymphocytes with highly specialized functions have been characterized. Some lymphocytes promote inflammation, while others have anti-inflammatory roles, and an optimal balance between these two opposing sets of lymphocytes is critical for immune homeostasis. A pro-inflammatory subset of CD4+ T helper 1 (Th1) lymphocytes known as cluster of differentiation 4 positive 28 negative T helper lymphocytes (CD4+CD28 null T cells) because they characteristically lack CD28 which is a co-stimulatory receptor critical for the activation and function of T cells.CD4+CD28 null T cells are rare in healthy individuals, but they increase in inflammatory and immune-mediated diseases. Prevalence of CD4+CD28 null T cells is high in chronic inflammatory diseases, autoimmune diseases, immunodeficiency and specific infectious diseases.It remains controversial whether CD4+CD28null T cells are antigen specific and which are the precise antigens that trigger their expansion. It has been suggested that CD4+CD28null T lymphocytes are auto-reactive and that repeated stimulation by auto-antigens drives the expansion of this cell subset.Expansion of the CD4+CD28 null T-cell subset in patients affected by autoimmune disorders has been linked to the severity of disease and an unfavourable prognosis.

ELIGIBILITY:
Inclusion Criteria:

* 1- newly diagnosed patients with AIHA 2- patients with idiopathic or secondary AIHA

Exclusion Criteria:

* 1-current steroid therapy 2- other concurrent chronic inflammatory conditions 3-recent blood transfusion 4- active Hepatitis C virus

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All newly diagnosed patients with AIHA without taking current steroid therapy ,other concurrent chronic inflammatory conditions ,recent blood transfusion or active Hepatitis C virus
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2023-01-30 (Estimated); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Role of CD4+CD28 null T helper lymphocytes in monitoring response to therapy in AIHA using flowcytometry in serum of AIHA patients. | Baseline
  The potential role of CD4+CD28 null T lymphocytes in monitoring response to therapy in AIHA .
  the percentage of circulating CD4+CD28 null T helper lymphocytes in AIHA either Idiopathic or Secondary using flowcytometry in serum of AIHA patients.

REFERENCES:
- [Background] Barcellini W. New Insights in the Pathogenesis of Autoimmune Hemolytic Anemia. Transfus Med Hemother. 2015 Sep;42(5):287-93. doi: 10.1159/000439002. Epub 2015 Sep 7. PMID 26696796
- [Background] Youssef SR, Elsalakawy WA. First report of expansion of CD4+/CD28 null T-helper lymphocytes in adult patients with idiopathic autoimmune hemolytic anemia. Hematol Transfus Cell Ther. 2021 Oct-Dec;43(4):396-401. doi: 10.1016/j.htct.2020.04.010. Epub 2020 Jul 16. PMID 32709527
- [Background] Fattizzo B, Barcellini W. Autoimmune Cytopenias in Chronic Lymphocytic Leukemia: Focus on Molecular Aspects. Front Oncol. 2020 Jan 10;9:1435. doi: 10.3389/fonc.2019.01435. eCollection 2019. PMID 31998632
- [Background] Jager U, Barcellini W, Broome CM, Gertz MA, Hill A, Hill QA, Jilma B, Kuter DJ, Michel M, Montillo M, Roth A, Zeerleder SS, Berentsen S. Diagnosis and treatment of autoimmune hemolytic anemia in adults: Recommendations from the First International Consensus Meeting. Blood Rev. 2020 May;41:100648. doi: 10.1016/j.blre.2019.100648. Epub 2019 Dec 5. PMID 31839434
- [Background] Broux B, Markovic-Plese S, Stinissen P, Hellings N. Pathogenic features of CD4+CD28- T cells in immune disorders. Trends Mol Med. 2012 Aug;18(8):446-53. doi: 10.1016/j.molmed.2012.06.003. Epub 2012 Jul 10. PMID 22784556
- [Background] Thewissen M, Somers V, Hellings N, Fraussen J, Damoiseaux J, Stinissen P. CD4+CD28null T cells in autoimmune disease: pathogenic features and decreased susceptibility to immunoregulation. J Immunol. 2007 Nov 15;179(10):6514-23. doi: 10.4049/jimmunol.179.10.6514. PMID 17982040